CLINICAL TRIAL: NCT07134920
Title: BCL6 Positivity and ART Outcomes: Comparing Norethindrone Acetate and Depo Lupron for Endometriosis Suppression Prior to Embryo Transfer
Brief Title: Norethindrone Impact on Receptiva Outcomes
Acronym: NIRO
Status: Active, not recruiting | Type: Observational
Sponsor: Inception Fertility Research Institute, LLC (Industry)
Collaborators: Cicero Diagnostic (Unknown)
Responsible Party: Sponsor
Other Study IDs: IRI-MLF-2025-002
Record Dates: First submitted 2025-08-14; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Infertility (IVF Patients); Infertility Female
Keywords: Receptiva; Depo Lupron Acetate; Norethindrone Acetate
MeSH Terms: conditions — Infertility; Infertility, Female

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Norethindrone acetate Group: Patients who received 6 and 8 weeks of suppression with norethindrone acetate prior to embryo transfer cycle
- Depo Leuprolide Group: Patients who received two monthly injections of Depo Leuprolide Acetate prior to embryo transfer cycle

SUMMARY:
This retrospective study aims to evaluate pregnancy outcomes in patients with a positive BCL6 test (ReceptivaDx, who were treated with either norethindrone acetate or Depo Lupron prior to embryo transfer. The current standard of care involves treatment with Depo Lupron, a GnRH agonist associated with significant hypoestrogenic side effects that mimic menopausal symptoms. Additionally, Depo Lupron is costly, with a retail price exceeding $2,000 per dose. In contrast, norethindrone acetate is a well-tolerated oral progestin, available at a fraction of the cost (under $100 for a one-month course). While prior studies have demonstrated comparable efficacy between Depo Lupron and norethindrone for managing endometriosis-associated pain, their relative effectiveness in improving reproductive outcomes-particularly in BCL6-positive patients undergoing embryo transfer-remains underexplored. This study seeks to address that gap by comparing ongoing pregnancy, live birth, and miscarriage rates between the two treatment groups.

Hypothesis: IVF Patients testing positive for BCL6 and treated with norethindrone will not do worse than the current recommended treatment of 60 days Depo leuprolide as defined by two endpoint metrics, pregnancy rate and live birth rate.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of recurrent pregnancy loss, recurrent implantation failure, unexplained infertility or severe dysmenorrhea and a positive BCL6 test Receptivadx
* Underwent assisted reproductive technology (ART or IVF)
* Treated with norethinedrone acetate 5 mg daily for 6 and 8 weeks or two monthly injections of Depo Leuprolide Acetate 7.5mg rior to embryo transfer cycle
* Euploid embryo transfer cycle was initiated within 1 week of completion of suppression protocol
* Adequate clinical documentation available, including treatment protocol, BCL6 results, and pregnancy outcomes
* If Endometrial Receptivity Analysis (ERA) was performed, result must be "receptive"
* A minimum uterine lining of 7.5mm was documented by ultrasound prior to the initiation of progesterone

Exclusion Criteria:

* Use of both norethinedrone acetate and Depo Leuprolide Acetate in the same treatment cycle
* Incomplete ART or outcome data
* Gestational carrier or egg donor
* No prescribed adjuvant therapy (e.g., Lovenox, Neupogen, IVIG)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women with a ReceptivaDx BCL6-positive test who completed hormonal suppression therapy prior to embryo transfer cycle
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2025-08-12 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Ongoing pregnancy rate | From beginning of treatment to 12 weeks post embryo transfer
  To compare ongoing pregnancy rates in BCL6-positive patients treated with norethindrone acetate versus Depo Lupron acetate

SECONDARY OUTCOMES:
Live birth rate | From start of treatment to 10 months post embryo transfer
  To compare live birth rates in BCL6-positive patients treated with norethindrone acetate versus Depo Lupron acetate
Miscarriage Rate | From start of treatment to 20 weeks post embryo transfer
  Defined as the loss of a clinically confirmed pregnancy before 20 weeks of gestation
Biochemical pregnancy rate | From start of treatment to 4 weeks post embryo transfer
  Defined as a low positive serum HCG with an inappropriate rise, spontaneous resolution
Ectopic pregnancy rate | From start of treatment to 8 weeks post embryo transfer

CONTACTS AND LOCATIONS:
Locations (1):
- Main Line Fertility, Bryn Mawr, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No